CLINICAL TRIAL: NCT00688051
Title: Changes in Adherence to Diet, Treatment and Medication in the Cystic Fibrosis Patient as a Result of Participation in a Simulation Game.
Brief Title: Changes in Adherence After Playing "My Life With CF" Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Craig A. Friesen, MD, Pediatric Gastroenterologist, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07 06-091E
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Adherence to treatment
MeSH Terms: conditions — Cystic Fibrosis; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: My Life with CF game

INTERVENTIONS:
Other: My Life with CF game — Play the game My Life with CF
  Other Names: My Life with CF

SUMMARY:
Nonadherence to treatment regimes among patients with cystic fibrosis (CF) is well documented in the literature. Unfortunately, few interventions have been successful at improving adherence rates in this patient population. Within the pediatric population, specifically adolescents, attitude toward treatment directly effects adherence to treatment. Changing attitude includes making conscious decisions regarding adherence or non-adherence and should include an understanding of what outcomes will likely result from nonadherence.

This study will determine if attitudes can be enhanced and adherence to treatment regimen improved in Cystic Fibrosis (CF) adolescent patients by using a simulation game "My Life with CF" . The target population is CF patients ages 12-21 years. Attitudes will be assessed utilizing four attitude scales in CF adolescents pre and post experiencing the simulation game. In the simulation game, patients make life decisions, including CF therapy decisions, using a fictional character diagnosed with CF. The game has been designed to help players understand the long-term effects of health care choices. Data from this pilot study will assess changes in attitudes and reported changes in adherence.

DETAILED DESCRIPTION:
Thirty patients will be enrolled in the study. These volunteer individuals will complete the Attitude Assessment Scale and Diet and Treatment form, play the game and provide demographic data. They will complete the Attitude Assessment Scales again following the game and debriefing. These individuals will complete the Attitude Assessment Scale and Diet and Treatment form a third time, one month after playing the game. Historical review indicates that enrollment for the study can be completed within 10 months after IRB approval is secured. This allows all aspects of the study to be complete within the one year time frame established by the funding agency.

Participants for this study will be identified using study inclusion / exclusion criteria Inclusion criteria are: 1) patients with a diagnosis of CF, 2) age 12 - 20 years, 3) capable of reading and conversing in English, 4) capable and willing to provide assent for study participation, and 5) presence of a parent/guardian capable of providing informed consent. Exclusion criteria are: 1) absence of a parent/guardian or unwillingness to provide permission, 2) potential participant declines to provide assent 3) the presence of a healthcare condition that does not meet infection control standards (i.e. patients with burkodalia cepacia) for participation in the small group setting necessary to play the game. Patients with MRSA will not be excluded from the study. Patients with MRSA can play the game alone, with a CMH staff member, study personnel, or sibling. All infection control measures will be followed according to hospital policy. Members of the study team have identified patients, based on inclusion criteria, who will qualify for the study. A letter will be mailed to these patients with a description of the game, study purpose, and time requirement. A follow-up phone call will be made by a member of the study team to arrange a time when the patient can play the game. Any questions related to study participation will be answered. Consent/assent will be obtained prior to filling out the paper work at the start of the game session.

When a patient is identified for study inclusion, a study investigator will explain the study to the parent/legal guardian and the child. If both these individuals express a willingness to participate, a copy of the informed consent/assent form will be given to them. After both the parent/guardian and child have read and signed the consent/assent form, a copy will be given to each of them and placed in the medical record. The original informed consent/assent form will be kept by the PI with all study materials. The study uses a convenience sampling methodology so no unique study number will be used.

3. Treatment Groups

There are no treatment groups for this study. Participants will complete an Attitude Assessment Scale and Diet and Treatment form prior to playing the game and complete the Attitude Assessment Scales immediately after the game and debriefing. The Attitude Assessment Scales and Diet and Treatment form will also be filled out again one month after playing the game. In addition, these individuals will provide self-disclosed demographic data, which will be used only to describe the study population.

4. Drugs/Devices/Experimental Intervention:

The experimental intervention includes playing the game "My Life with CF."

Each participant will complete an assessment regarding diet and treatment adherence, and attitudes toward behaviors associated with 1) belief that luck rather than effort determines what happens to a person in life, 2) belief in personal invulnerability, and 3) making life decisions without including long-term consequences. After the baseline measure has been obtained, participants will play the "My Life with CF" game. The attitude assessment scales will be repeated after the game and debriefing. The attitude assessment scales and Diet and Treatment form will be repeated one month following the game.

5. Observations and Measurements

Participants will be asked to complete the "Attitude Assessment Scales provided in Appendix B. Attitude Scales 1,2 and 3 are the attitude scales validated for the "My Life" game. Attitude scale 4 was created specifically for the "My Life with CF" game and has not been validated. Each attitude scale has 20 questions and is based on a likert-type scale with 1 strongly disagree to 5 strongly agree. The first three attitude scales focus on the three attitudes which have been shown to influence decision making during adolescence. Attitude scale number one assesses personal invulnerability, attitude scale number two assesses present versus future considerations, and attitude scale number three measures luck versus effort. Attitude scale number 4 has an equal number of questions from the above three categories which are specific to CF.

Data collection will occur through the utilization of a "My Life with CF" Case Report Form provided in Appendix C. All study participants' personal health information will be kept confidential in compliance with Federal Law and institutional guidelines. All research case report forms will be kept in Kathy Christenson's office within a secured cabinet and destroyed in accordance with policy and procedures in place regarding research data.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a diagnosis of CF
2. age 12 - 20 years
3. capable of reading and conversing in English
4. capable and willing to provide assent for study participation
5. presence of a parent/guardian capable of providing informed consent

Exclusion Criteria:

1. absence of a parent/guardian or unwillingness to provide permission
2. potential participant declines to provide assent
3. the presence of a healthcare condition that does not meet infection control standards (i.e. patients with burkodalia cepacia) for participation in the small group setting necessary to play the game.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine changes in attitude associated with playing the game "My Life with CF". | One month follow up

SECONDARY OUTCOMES:
To determine changes in frequency to adherence of treatment plan, specifically related to respiratory treatments and medications, one month after playing the game "My Life with CF". | One month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Christenson, RN CPNP, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States